CLINICAL TRIAL: NCT06090747
Title: Efecto de Una intervención Multidisciplinaria de Estilo de Vida Sobre el Exposoma de Pacientes premenopáusicas Con cáncer de Mama Estadios I-III.
Brief Title: Improving Lifestyle Behavior by "Joven, Fuerte y Saludable" Multidisciplinary Program.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: Anahuac University (Other); Tecnologico de Monterrey (Other); Instituto Nacional de Rehabilitacion (Other Government); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Marlid Cruz Ramos, PhD, Instituto Nacional de Cancerologia de Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 023-005-OMI(CEI-05022)
Record Dates: First submitted 2023-09-07; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasm
Keywords: Multidisciplinary; Intervention; Lifestyle; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A controlled trial design was adopted in which patients were assigned to two intervention groups according to the nutritional, psychological, or rehabilitation risk at baseline or according to their geographical localization. The first group will receive a hybrid multidisciplinary lifestyle education intervention (control), whereas the second group will receive an individualized hybrid multidisciplinary lifestyle intervention. The study aims to evaluate the effect of both interventions on the internal exposome of young patients with breast cancer and their effect on quality of life. To do this, changes over time in biochemical, inflammatory, and metabolomic indicators will be measured, and validated questionnaires will be applied to assess lifestyle components such as level of physical activity, sleep hygiene, emotional distress, and quality of life (so baseline, during and after treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluate the effect of hybrid educational intervention in Lifestyle behavior. (Active Comparator): Group 1: hybrid educational intervention
  Interventions: Behavioral: Hybrid lifestyle educational multidisciplinary intervention.
- Evaluate the effect of hybrid personalized intervention in Lifestyle behavior (Experimental): Group 2: hybrid personalized lifestyle intervention delivered by a multidisciplinary team of specialists in oncology, nutrition, psychology, rehabilitation and mindfulness.
  Interventions: Behavioral: Hybrid lifestyle personalized multidisciplinary intervention.

INTERVENTIONS:
Behavioral: Hybrid lifestyle educational multidisciplinary intervention. — Participants will receive a standardized educational healthy lifestyle intervention. The information will be shared via digital tools such as mail, WhatsApp, zoom workshops, educational videos, "Joven, Fuerte y Saludable" webpage, "Joven, Fuerte y Saludable" mobile app, and face-to-face educational sessions.
  Arms: Evaluate the effect of hybrid educational intervention in Lifestyle behavior.
Behavioral: Hybrid lifestyle personalized multidisciplinary intervention. — Participants will receive a standardized educational healthy lifestyle intervention and personalized lifestyle intervention based on their clinical evaluation. Based on clinical records participants will be sent to nutritional, psychological, rehabilitation, and Mindfulness intervention. Educational and motivational strategies include digital tools such as mail, WhatsApp, zoom workshops, educational videos, the "Joven, Fuerte y Saludable" webpage, and the "Joven, Fuerte y Saludable" mobile app. And individualized follow-up through Mobile apps such as AVENA
  Arms: Evaluate the effect of hybrid personalized intervention in Lifestyle behavior

SUMMARY:
Breast cancer is the leading cause of mortality in women worldwide. Latin-American women are diagnosed at younger ages, in advanced stages, and with aggressive molecular subtypes. Lifestyle seems related to these aggressive conditions and worse outcomes. The present study seeks to evaluate the effect of a hybrid multidisciplinary intervention for implementing a healthy lifestyle to modify the personal and internal exposome of young women with breast cancer. This randomized controlled experimental study with two groups:

Group 1: Hybrid multidisciplinary lifestyle education intervention. Group 2: Individualized hybrid multidisciplinary lifestyle interventions. The multidisciplinary lifestyle intervention program includes oncology, nutrition, physiotherapy, and psychology interventions.

DETAILED DESCRIPTION:
Breast cancer (BC) is a leading cause of death in women worldwide, especially in Latin America, where patients often present with advanced stages of aggressive subtypes of BC at a younger age. The risk of BC depends on various factors, including hormone replacement therapy history, reproductive history, alcohol or tobacco consumption, physical activity, and dietary habits, collectively called exposome. Exposome refers to the exposure to environmental influences and biological responses throughout a person's life from the prenatal stage. It can be influenced by the environment, diet, behavior, and endogenous processes.

External exposome refers to environmental factors such as mental stress, climate, and lifestyle. In contrast, internal exposome are changes within an organism, such as increased stress hormones, inflammatory cytokines, and oxidative stress. Constant exposure to environmental factors, such as an unhealthy lifestyle, can cause cellular damage and contribute to the growth and evolution of tumors. Once cellular damage occurs, internal exposome promotes changes that create a harmful environment, favoring cancer cells to acquire coping mechanisms for stress and drugs, leading to resistance to oncological treatments.

Obesity is part of the personal exposome and can impact the internal exposome, potentially affecting BC patients. A significant percentage of patients diagnosed with BC (70.9%) are overweight or obese at the time of diagnosis. This weight gain usually occurs during systemic treatment, with 25% of patients gaining weight within six months, 32% between 6-12 months, and 20% between 12-18 months after diagnosis. Young women with breast cancer (YWBC) also experience an increase in weight since the initiation of oncological treatment and up to the second year of diagnosis (from 39% at baseline to 46% in two years), highlighting the importance of evaluating the implications of weight gain and whether early intervention would help control the risk factors mentioned earlier. Obesity may also be associated with worse disease-free and overall survival.

Weight gain in patients with BC is often associated with several factors, including systemic treatment, diagnosis at a young age, and lifestyle changes resulting from the disease or treatment. However, reduced physical activity is the primary mechanism underlying weight gain. The combination of chemotherapy and endocrine therapy is linked to higher weight gain, especially in patients who are premenopausal (an increase of up to 24 kg). In contrast, postmenopausal women tend to lose weight.

BC patients have reported experiencing physical symptoms and psychological distress, which can negatively impact their quality of life (QoL). These symptoms can affect their physical functioning, psychological well-being, and social support levels. YWBC is a vulnerable population with specific concerns such as fertility, self-image, QoL, sexuality, and personal goals and experience high anxiety and depression. Maintaining a healthy lifestyle can improve QoL and lead to better prognoses and lower mortality rates. For example, exercise can reduce breast cancer-related death risk by 30% and all-cause death risk by 41%. Patients undergoing oncology treatment face various nutritional challenges that differ based on the type and stage of cancer, and the treatments may worsen these challenges. Early nutritional screening and interventions are crucial in the cancer population, as emphasized in the clinical guidelines (ASPEN/ESPEN).

The Instituto Nacional de Cancerología (INCAN) in Mexico City offers a program called "Joven & Fuerte" for young women diagnosed with BC. However, the attention was not systematic, and it was difficult to measure the benefits of the intervention. So, the present study proposes a psychological intervention, side effect management, physical activity, sleep hygiene, and psychological strategies, with onsite and remote interventions to improve patient adherence and ensure timely attention. The study aims to evaluate the impact of early intervention on metabolic control in newly diagnosed BC patients, their QoL, and clinical outcomes.

METHODS A controlled trial design was adopted in which patients were assigned to two intervention groups according to the nutritional, psychological, or rehabilitation risk at baseline or according to their geographical localization. The first group will receive a hybrid multidisciplinary lifestyle education intervention, whereas the second group will receive an individualized hybrid multidisciplinary lifestyle intervention.

Patients will be recruited through an active program at the INCAN, where potential candidates will be identified and invited by the navigator at the program "Joven & Fuerte." After they sign the informed consent form (ICF), patients will be assigned into one of the two groups:

Group 1: Hybrid multidisciplinary lifestyle education intervention. Group 2: Individualized hybrid multidisciplinary lifestyle interventions. The initial proposal was a randomized assignment to each group; however, the pilot study revealed challenges for patients who lived far from the hospital, in other states or had personal obligations such as family or work. Therefore, the randomization process was adapted to meet the patient's needs. The intervention aims to facilitate patients' adherence and follow-up with healthcare providers. Additionally, patient preferences were considered when assigning them to a group.

Objectives.

To assess the ability of a personalized lifestyle intervention to support breast cancer patients undergoing active treatment to maintain or obtain a healthy lifestyle.

To evaluate adopting a healthy lifestyle, validated questionnaires will be applied to assess lifestyle components such as level of physical activity, sleep hygiene, and emotional distress (baseline, during, and after treatment).

To evaluate changes in internal exposome parameters such as body composition, biochemical, inflammatory, and metabolomic indicators will be measured.

To evaluate the effectiveness of a virtual educational program to support breast cancer patients in active treatment to maintain or obtain a healthy personal exposome and its usefulness in patients who live in remote locations or cannot attend a face-to-face consultation.

To evaluate the motivational and educational effect of a personalized follow-up by phone, Zoom, WhatsApp, or social networks.

To evaluate the implementation's effect on participants' quality of life. To evaluate the barriers and challenges to implementing the healthy life intervention.

The proposed indicators will make it possible to measure the effect of the proposed intervention on the exposome of the patients, as well as adherence to the intervention, through attendance at consultations and changes in lifestyle using validated questionnaires. Among the interventions, an individualized hybrid format is proposed, both with face-to-face consultations, as well as remote follow-up through telephone calls, video calls, or material sent through digital platforms, which will benefit patients who are far from the institute or who they have difficulties to attend due to travel times, work schedules; which translates into greater adherence to the intervention and positive changes in the lifestyle of patients. Finally, it is proposed to produce an educational manual and other printed or video support materials for patients, allowing the program to be replicated in other centers with similar needs in Mexico and Latin America. Additionally, the present study intends to use the variables obtained: the clinical, anthropometric, biochemical, inflammatory profile, and metabolites identified as possible biomarkers to develop a predictor algorithm for the deterioration of quality of life in patients.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with stage I-III BC, confirmed by pathology and image at the INCAN
* Candidates for multidisciplinary treatment including surgery, chemotherapy, and/or hormonal treatments.
* Signed the informed consent form
* Have access to a mobile phone or any electronic device with an active internet connection to receive the program information.

Exclusion Criteria:

* Patients with inflammatory cancer
* Those with cardiomyopathy or ventricular dysfunction (NYHA >II), arrythmia secondary to left ventricular ejection alterations that requires medication, previous myocardial infarction, or angina pectoris in the last six months
* Receiving treatment for cardiovascular or cerebrovascular disease, inflammatory bowel disease, malabsorption syndrome, rheumatoid arthritis, lupus, thyroid diseases, or Cushing syndrome
* Unable to walk for at least 1 km
* Have cardiovascular, respiratory, or musculoskeletal diseases that impede physical activity
* Pregnant or breastfeeding
* Have psychiatric conditions impeding active participation in this protocol
* Do not understand Spanish

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adoption of healthy lifestyle | Baseline evaluation and final evaluation (18 months).
  The patient lifestyle compliance measured by the scores of World Cancer Research Fund (WCRF) / American Institute for Cancer Research (AICR) questionnaire, SCORE ≥ 5
Changes on 24-hour reminder | Baseline, 3, 6, 12 and 18 months.
  Evaluate the changes on daily nutritional intake (total energy, carbohydrate, protein and, lipids grams)
Education and Motivational effectiveness of digital tools. | 3, 6, 12 and 18 months.
  To evaluate the motivational and educational effect of a personalized follow-up by phone, Zoom, WhatsApp, or social networks (number of views in videos, number of Zoom sessions, number o WA calls).
Physical Activity changes | Baseline, 3, 6,12 and 18 months.
  Evaluate the changes on physical activitiy by International Physical Activity Questionnaire (IPAQ) score (high: 1500 to 3000 METS per/week; moderate: 600 MET per/week.
Quality of sleep changes | Baseline, 3, 6,12 and 18 months.
  Evaluate the quality of sleep changes by Pittsburgh Sleep Quality Index (PSQI). Total Score 0 to 21. Score 0 (No sleep difficulty); Score 1 to7 (mild sleep difficulty); Score 8-14 (moderate sleep dificulty); 15-21 (severe sleep difficulty).
Depression risk evaluation | Baseline, 3, 6,12 and 18 months.
  Patient Health Questionnaire (PHQ-9) 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
Anxiety risk evaluation | Baseline, 3, 6,12 and 18 months.
  Generalized Anxiety Disorder Assessment (GAD-7) 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Minfulness evaluation - How having a concentrated mind affects on daily life | Baseline, 3, 6,12 and 18 months.
  Five Facet Mindfulness Questionnaire (FFMQ) 1-2: Lack of concentrated mind 3: Intermediate attention awareness 4-5: Advance attention awareness
Body composition - Body fat | Baseline, 3, 6,12 and 18 months.
  To evaluate the Effect of lifestyle intervention on:
  Body fat percentage (acceptable fat percentage <31%)
Biochemical parameters - Inflammatory cytokines | Baseline, 3, 6,12 and 18 months.
  To evaluate the effect of lifestyle intervention on biochemical parameters:
  Cytokines level
Anthropometric measurements - Body weight | Baseline, 3, 6,12 and 18 months.
  Changes in:
  Body weight (kg)
Minfulness evaluation - Disposition to attention awareness | Baseline, 3, 6,12 and 18 months.
  Mindful Attention Awareness Scale (MAAS) 1-2: Lack of attention awareness 3: Intermediate attention awareness 4-5: Advance attention awareness 6: Overvalued (questionnaire was notanswered honestly)
Minfulness evaluation - Disposition to mindfulness | Baseline, 3, 6,12 and 18 months.
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) 1-2: Lack of disposition 3: Intermediate disposition 4: Advance into mindfulness
Body composition - Muscle | Baseline, 3, 6,12 and 18 months.
  To evaluate the Effect of lifestyle intervention on:
  Muscle (muscle mass in kg and muscle mass index ≤6.42 kg/m2)
Biochemical parameters - Glucose | Baseline, 3, 6,12 and 18 months.
  To evaluate the effect of lifestyle intervention on biochemical parameters:
  Blood glucose <135mg/dL
Biochemical parameters - Lipid profile | Baseline, 3, 6,12 and 18 months.
  To evaluate the effect of lifestyle intervention on biochemical parameters:
  LDL<100mg/dL, HDL >40mg/dL and triglycerides <150mg/dL)
Anthropometric measurements - Waist circumference | Baseline, 3, 6,12 and 18 months.
  Changes in:
  Waist circumference (cm)
Anthropometric measurements - Waist to hip ratio | Baseline, 3, 6,12 and 18 months.
  Changes in:
  Waist to hip ratio (<0.8)

SECONDARY OUTCOMES:
Improvement of quality of life parameters with lifestyle intervention- QLQ-C30 | Baseline, 3, 6 ,12 and 18 months.
  Effect of lifestyle intervention on quality of life measured by European Organization of Research and Treatment of Cancer Quality of Life Questionnarie (QLQ-C30)
Barriers and challenges to implement the lifestyle intervention - CFIR | 3, 6, 12 and 18 months.
  To identify the barriers and challenges for the implementation of the healthy lifestyle intervention.
  CFIR (Consolidated Framework for Implementation Research) - qualitative evaluation
Barriers and challenges to implement the lifestyle intervention - RE-AIM | 3, 6, 12 and 18 months.
  To identify the barriers and challenges for the implementation of the healthy lifestyle intervention.
  RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance)
Improvement of quality of life parameters with lifestyle intervention- QLQ-BR23 | Baseline, 3, 6 ,12 and 18 months.
  Effect of lifestyle intervention on quality of life measured by Quality of Life Questionnarie Breast Cancer (QLQ-BR23) - Sympton scale score.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Marlid Cruz Ramos, México, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amadou A, Torres-Mejia G, Hainaut P, Romieu I. Breast cancer in Latin America: global burden, patterns, and risk factors. Salud Publica Mex. 2014 Sep-Oct;56(5):547-54. doi: 10.21149/spm.v56i5.7379. PMID 25604300
- [Background] Bessonneau V, Rudel RA. Mapping the Human Exposome to Uncover the Causes of Breast Cancer. Int J Environ Res Public Health. 2019 Dec 27;17(1):189. doi: 10.3390/ijerph17010189. PMID 31892107
- [Background] Fang M, Hu L, Chen D, Guo Y, Liu J, Lan C, Gong J, Wang B. Exposome in human health: Utopia or wonderland? Innovation (Camb). 2021 Oct 6;2(4):100172. doi: 10.1016/j.xinn.2021.100172. eCollection 2021 Nov 28. PMID 34746906
- [Background] Daiber A, Kroller-Schon S, Frenis K, Oelze M, Kalinovic S, Vujacic-Mirski K, Kuntic M, Bayo Jimenez MT, Helmstadter J, Steven S, Korac B, Munzel T. Environmental noise induces the release of stress hormones and inflammatory signaling molecules leading to oxidative stress and vascular dysfunction-Signatures of the internal exposome. Biofactors. 2019 Jul;45(4):495-506. doi: 10.1002/biof.1506. Epub 2019 Apr 2. PMID 30937979
- [Background] Kalita-de Croft P, Sharma S, Sobrevia L, Salomon C. Extracellular vesicle interactions with the external and internal exposome in mediating carcinogenesis. Mol Aspects Med. 2022 Oct;87:101039. doi: 10.1016/j.mam.2021.101039. Epub 2021 Oct 8. PMID 34629184
- [Background] Barquera S, Hernandez-Barrera L, Trejo-Valdivia B, Shamah T, Campos-Nonato I, Rivera-Dommarco J. [Obesity in Mexico, prevalence andtrends in adults. Ensanut 2018-19.]. Salud Publica Mex. 2020 Nov-Dec;62(6):682-692. doi: 10.21149/11630. Spanish. PMID 33620965
- [Background] Reynoso-Noveron N, Villarreal-Garza C, Soto-Perez-de-Celis E, Arce-Salinas C, Matus-Santos J, Ramirez-Ugalde MT, Alvarado-Miranda A, Cabrera-Galeana P, Meneses-Garcia A, Lara-Medina F, Bargallo-Rocha E, Mohar A. Clinical and Epidemiological Profile of Breast Cancer in Mexico: Results of the Seguro Popular. J Glob Oncol. 2017 Dec;3(6):757-764. doi: 10.1200/JGO.2016.007377. Epub 2017 Feb 8. PMID 29244990
- [Background] Villarreal-Garza C, Platas A, Miaja M, Fonseca A, Mesa-Chavez F, Garcia-Garcia M, Chapman JA, Lopez-Martinez EA, Pineda C, Mohar A, Galvez-Hernandez CL, Castro-Sanchez A, Martinez-Cannon BA, Barragan-Carrillo R, Munoz-Lozano JF, Goss P, Bargallo-Rocha JE, Aguilar D, Cardona S, Canavati M. Young Women With Breast Cancer in Mexico: Results of the Pilot Phase of the Joven & Fuerte Prospective Cohort. JCO Glob Oncol. 2020 Mar;6:395-406. doi: 10.1200/JGO.19.00264. PMID 32142405
- [Background] Shaikh H, Bradhurst P, Ma LX, Tan SYC, Egger SJ, Vardy JL. Body weight management in overweight and obese breast cancer survivors. Cochrane Database Syst Rev. 2020 Dec 11;12(12):CD012110. doi: 10.1002/14651858.CD012110.pub2. PMID 33305350
- [Background] Bustamante-Marin XM, Merlino JL, Devericks E, Carson MS, Hursting SD, Stewart DA. Mechanistic Targets and Nutritionally Relevant Intervention Strategies to Break Obesity-Breast Cancer Links. Front Endocrinol (Lausanne). 2021 Mar 17;12:632284. doi: 10.3389/fendo.2021.632284. eCollection 2021. PMID 33815289
- [Background] Villarreal-Garza C, Platas A, Miaja M, Mesa-Chavez F, Garcia-Garcia M, Fonseca A, Pineda C, de la Rosa-Pacheco S, Galvez-Hernandez CL, Bargallo-Rocha E, Castro J, Rodriguez-Gomez D, Cruz-Ramos M, Mohar A. Patients' satisfaction with a supportive care program for young breast cancer patients in Mexico: Joven & Fuerte supports patients' needs and eases their illness process. Support Care Cancer. 2020 Oct;28(10):4943-4951. doi: 10.1007/s00520-020-05334-y. Epub 2020 Feb 4. PMID 32020358
- [Background] Perry S, Kowalski TL, Chang CH. Quality of life assessment in women with breast cancer: benefits, acceptability and utilization. Health Qual Life Outcomes. 2007 May 2;5:24. doi: 10.1186/1477-7525-5-24. PMID 17474993
- [Background] Montagnese C, Porciello G, Vitale S, Palumbo E, Crispo A, Grimaldi M, Calabrese I, Pica R, Prete M, Falzone L, Libra M, Cubisino S, Poletto L, Martinuzzo V, Coluccia S, Esindi N, Nocerino F, Minopoli A, Grilli B, Fiorillo PC, Cuomo M, Cavalcanti E, Thomas G, Cianniello D, Pinto M, De Laurentiis M, Pacilio C, Rinaldo M, D'Aiuto M, Serraino D, Massarut S, Caggiari L, Evangelista C, Steffan A, Catalano F, Banna GL, Scandurra G, Ferrau F, Rossello R, Antonelli G, Guerra G, Farina A, Messina F, Riccardi G, Gatti D, Jenkins DJA, Celentano E, Botti G, Augustin LSA. Quality of Life in Women Diagnosed with Breast Cancer after a 12-Month Treatment of Lifestyle Modifications. Nutrients. 2020 Dec 31;13(1):136. doi: 10.3390/nu13010136. PMID 33396551
- [Background] Ruiz-Vozmediano J, Lohnchen S, Jurado L, Recio R, Rodriguez-Carrillo A, Lopez M, Mustieles V, Exposito M, Arroyo-Morales M, Fernandez MF. Influence of a Multidisciplinary Program of Diet, Exercise, and Mindfulness on the Quality of Life of Stage IIA-IIB Breast Cancer Survivors. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420924757. doi: 10.1177/1534735420924757. PMID 32462950
- [Background] Ee C, Cave A, Vaddiparthi V, Naidoo D, Boyages J. Factors associated with weight gain after breast cancer: Results from a community-based survey of Australian women. Breast. 2023 Jun;69:491-498. doi: 10.1016/j.breast.2023.01.012. Epub 2023 Jan 25. PMID 36710237
- [Background] Nyrop KA, Deal AM, Shachar SS, Park J, Choi SK, Lee JT, O'Hare EA, Wheless A, Carey LA, Muss HB. Weight trajectories in women receiving systemic adjuvant therapy for breast cancer. Breast Cancer Res Treat. 2020 Feb;179(3):709-720. doi: 10.1007/s10549-019-05501-8. Epub 2019 Nov 16. PMID 31734823
- [Background] Richards J, Arensberg MB, Thomas S, Kerr KW, Hegazi R, Bastasch M. Impact of Early Incorporation of Nutrition Interventions as a Component of Cancer Therapy in Adults: A Review. Nutrients. 2020 Nov 5;12(11):3403. doi: 10.3390/nu12113403. PMID 33167544
- [Background] Li YR, Ro V, Tchou JC. Obesity, Metabolic Syndrome, and Breast Cancer: From Prevention to Intervention. Curr Surg Rep. 2018 Mar;6(3):7. doi: 10.1007/s40137-018-0204-y. Epub 2018 Feb 24. PMID 31293823
- [Background] Cnop M, Foufelle F, Velloso LA. Endoplasmic reticulum stress, obesity and diabetes. Trends Mol Med. 2012 Jan;18(1):59-68. doi: 10.1016/j.molmed.2011.07.010. Epub 2011 Aug 31. PMID 21889406
- [Background] Bose S, Allen AE, Locasale JW. The Molecular Link from Diet to Cancer Cell Metabolism. Mol Cell. 2020 Jun 18;78(6):1034-1044. doi: 10.1016/j.molcel.2020.05.018. Epub 2020 Jun 5. PMID 32504556
- [Background] De Cicco P, Catani MV, Gasperi V, Sibilano M, Quaglietta M, Savini I. Nutrition and Breast Cancer: A Literature Review on Prevention, Treatment and Recurrence. Nutrients. 2019 Jul 3;11(7):1514. doi: 10.3390/nu11071514. PMID 31277273
- [Background] Hoy MK, Winters BL, Chlebowski RT, Papoutsakis C, Shapiro A, Lubin MP, Thomson CA, Grosvenor MB, Copeland T, Falk E, Day K, Blackburn GL. Implementing a low-fat eating plan in the Women's Intervention Nutrition Study. J Am Diet Assoc. 2009 Apr;109(4):688-96. doi: 10.1016/j.jada.2008.12.016. PMID 19328264
- [Background] Demark-Wahnefried W, Hars V, Conaway MR, Havlin K, Rimer BK, McElveen G, Winer EP. Reduced rates of metabolism and decreased physical activity in breast cancer patients receiving adjuvant chemotherapy. Am J Clin Nutr. 1997 May;65(5):1495-501. doi: 10.1093/ajcn/65.5.1495. PMID 9129482
- [Background] Makari-Judson G, Braun B, Jerry DJ, Mertens WC. Weight gain following breast cancer diagnosis: Implication and proposed mechanisms. World J Clin Oncol. 2014 Aug 10;5(3):272-82. doi: 10.5306/wjco.v5.i3.272. PMID 25114844
- [Background] KABAT-ZINN, Jon. Mindfulness-based interventions in context: past, present, and future. 2003.
- [Background] Villarreal-Garza C, Aguila C, Platas A, Lara-Guerra H. [Clinical Forum: Breast cancer in young women in Mexico: unmet needs and clinical challenges]. Rev Invest Clin. 2014 Nov-Dec;66(6):547-58. No abstract available. Spanish. PMID 25729872
- [Background] Campbell-Enns H, Woodgate R. The psychosocial experiences of women with breast cancer across the lifespan: a systematic review protocol. JBI Database System Rev Implement Rep. 2015 Jan;13(1):112-21. doi: 10.11124/jbisrir-2015-1795. PMID 26447012
- [Background] Gálvez-Hernández CL, Ortega Mondragón A, Villarreal-Garza C, Ramos Del Río B. Young women with breast cancer: Supportive care needs and resilience. Psicooncologia (Pozuelo de Alarcon). 2018;15(2):287-300.
- [Background] Guarino A, Polini C, Forte G, Favieri F, Boncompagni I, Casagrande M. The Effectiveness of Psychological Treatments in Women with Breast Cancer: A Systematic Review and Meta-Analysis. J Clin Med. 2020 Jan 12;9(1):209. doi: 10.3390/jcm9010209. PMID 31940942
- [Background] Lengacher CA, Reich RR, Paterson CL, Shelton M, Shivers S, Ramesar S, Pleasant ML, Budhrani-Shani P, Groer M, Post-White J, Johnson-Mallard V, Kane B, Cousin L, Moscoso MS, Romershausen TA, Park JY. A Large Randomized Trial: Effects of Mindfulness-Based Stress Reduction (MBSR) for Breast Cancer (BC) Survivors on Salivary Cortisol and IL-6. Biol Res Nurs. 2019 Jan;21(1):39-49. doi: 10.1177/1099800418789777. Epub 2018 Aug 5. PMID 30079756
- [Background] Widiasih R, Ermiati, Jayanti TN, Rais Y. Psychosocial Interventions for Improving the Quality of Life in Breast Cancer Survivors: A Literature Review. In: IOP Conference Series: Earth and Environmental Science. Institute of Physics Publishing; 2019.
- [Background] Rogers LQ, Courneya KS, Oster RA, Anton PM, Robbs RS, Forero A, McAuley E. Physical Activity and Sleep Quality in Breast Cancer Survivors: A Randomized Trial. Med Sci Sports Exerc. 2017 Oct;49(10):2009-2015. doi: 10.1249/MSS.0000000000001327. PMID 28538261
- [Background] Urech C, Grossert A, Alder J, Scherer S, Handschin B, Kasenda B, Borislavova B, Degen S, Erb J, Faessler A, Gattlen L, Schibli S, Werndli C, Gaab J, Berger T, Zumbrunn T, Hess V. Web-Based Stress Management for Newly Diagnosed Patients With Cancer (STREAM): A Randomized, Wait-List Controlled Intervention Study. J Clin Oncol. 2018 Mar 10;36(8):780-788. doi: 10.1200/JCO.2017.74.8491. Epub 2018 Jan 25. PMID 29369731
- [Background] van den Berg SW, Gielissen MF, Custers JA, van der Graaf WT, Ottevanger PB, Prins JB. BREATH: Web-Based Self-Management for Psychological Adjustment After Primary Breast Cancer--Results of a Multicenter Randomized Controlled Trial. J Clin Oncol. 2015 Sep 1;33(25):2763-71. doi: 10.1200/JCO.2013.54.9386. Epub 2015 Jul 13. PMID 26169621
- [Background] Dieli-Conwright CM, Wong L, Waliany S, Bernstein L, Salehian B, Mortimer JE. An observational study to examine changes in metabolic syndrome components in patients with breast cancer receiving neoadjuvant or adjuvant chemotherapy. Cancer. 2016 Sep 1;122(17):2646-53. doi: 10.1002/cncr.30104. Epub 2016 May 24. PMID 27219902
- [Background] Snetselaar LG, de Jesus JM, DeSilva DM, Stoody EE. Dietary Guidelines for Americans, 2020-2025: Understanding the Scientific Process, Guidelines, and Key Recommendations. Nutr Today. 2021 Nov-Dec;56(6):287-295. doi: 10.1097/NT.0000000000000512. Epub 2021 Nov 12. PMID 34987271
- [Background] Fowler S. Diabetes Prevention Program (V8) . NIDDK Central Repository. 2023; Resources for Research (R4R), https://repository.niddk.nih.gov/.
- [Background] Hauner D, Rack B, Friedl T, Hepp P, Janni W, Hauner H. Rationale and description of a lifestyle intervention programme to achieve moderate weight loss in women with non-metastatic breast cancer: the lifestyle intervention part of the SUCCESS C Study. BMJ Nutr Prev Health. 2020 Sep 21;3(2):213-219. doi: 10.1136/bmjnph-2020-000119. eCollection 2020 Dec. PMID 33521531
- [Background] Di Meglio A, Martin E, Crane TE, Charles C, Barbier A, Raynard B, Mangin A, Tredan O, Bouleuc C, Cottu PH, Vanlemmens L, Segura-Djezzar C, Lesur A, Pistilli B, Joly F, Ginsbourger T, Coquet B, Pauporte I, Jacob G, Sirven A, Bonastre J, Ligibel JA, Michiels S, Vaz-Luis I. A phase III randomized trial of weight loss to reduce cancer-related fatigue among overweight and obese breast cancer patients: MEDEA Study design. Trials. 2022 Mar 4;23(1):193. doi: 10.1186/s13063-022-06090-6. PMID 35246219
- [Background] Febvey-Combes O, Jobard E, Rossary A, Pialoux V, Foucaut AM, Morelle M, Delrieu L, Martin A, Caldefie-Chezet F, Touillaud M, Berthouze SE, Boumaza H, Elena-Herrmann B, Bachmann P, Tredan O, Vasson MP, Fervers B. Effects of an Exercise and Nutritional Intervention on Circulating Biomarkers and Metabolomic Profiling During Adjuvant Treatment for Localized Breast Cancer: Results From the PASAPAS Feasibility Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:1534735420977666. doi: 10.1177/1534735420977666. PMID 33655799

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT06090747/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT06090747/ICF_001.pdf